CLINICAL TRIAL: NCT07348523
Title: Comparison of the Effectiveness of Classical and Modified Erector Spinae Plane Blocks in Postoperative Analgesia Management Following Lumbar Spinal Surgery: A Prospective Study
Brief Title: Comparison of the Postoperative Analgesic Efficacy of Classical and Modified Erector Spinae Plane Blocks After Lumbar Spinal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: OMUKAEK 2025/247
Record Dates: First submitted 2025-12-31; First posted 2026-01-16 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: Acute Pain; Spinal Stenosis Lumbar
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: Group K-ESP (Active Comparator): The erector spinae plane block will be performed 30 minutes before lumbar spine surgery.
  Interventions: Other: The Classical Erector Spinae Plane Block
- Active Comparator: Group M-ESP (Active Comparator): The modified erector spinae plane block will be performed 30 minutes before lumbar spine surgery.
  Interventions: Other: Modified Erector Spinae Plane Blocks

INTERVENTIONS:
Other: The Classical Erector Spinae Plane Block — The erector spinae plane block will be performed under ultrasound guidance before the induction of general anesthesia.
  Arms: Active Comparator: Group K-ESP
Other: Modified Erector Spinae Plane Blocks — Modified erector spinae plane blocks will be performed under ultrasound guidance before the induction of general anesthesia.
  Arms: Active Comparator: Group M-ESP

SUMMARY:
The investigators aim to compare the postoperative analgesic efficacy of the classical erector spinae plane block and the modified erector spinae plane block in the management of postoperative analgesia after lumbar disc surgery.

DETAILED DESCRIPTION:
Lumbar spinal stenosis may lead to variable signs and symptoms such as low back pain, radiating pain to the lower extremities, and reduced walking capacity. Lumbar disc surgery itself causes significant pain due to extensive dissection and muscle retraction during the procedure. A multimodal analgesic approach is preferred for postoperative pain management after lumbar spine surgery. The addition of regional anesthesia techniques reduces opioid-related side effects and is associated with earlier mobilization, shorter hospital stay, and improved patient satisfaction.

In patients undergoing lumbar disc surgery, the classical erector spinae plane block and the modified erector spinae plane block provide effective analgesia for postoperative pain control.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 years,
* Classified as ASA physical status I-III,
* Scheduled to undergo single-level lumbar spinal surgery under general anesthesia
* Who agree to participate in the study by providing written informed consent

Exclusion Criteria:

* History of bleeding diathesis or current anticoagulant therapy
* Known allergy or hypersensitivity to local anesthetics or opioid medications
* Infection at the planned block injection site
* Previous lumbar spine surgery
* History of gabapentinoid or corticosteroid use within the last 3 weeks
* Inability to use a patient-controlled analgesia (PCA) device
* Suspected pregnancy, confirmed pregnancy, or breastfeeding Refusal to undergo the procedure or to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | 24 hours
  In the postoperative period, patients will be given opioids according to their pain density with a patient-controlled device, and the daily Morphine consumption in Patient Controlled Analgesia device will be collected and compared between groups.

SECONDARY OUTCOMES:
Perioperative pain intensity | 24 hours
  Changes in the Numerical Rating Scale (NRS) will be recorded at rest and during movement. The participant's baseline NRS will be recorded, followed by measurements before and after neuraxial positioning and up to 24 hours post-surgery.
  The NRS is a unidimensional measure of pain intensity in adults. It is a segmented numerical version of the Visual Analog Scale (VAS) where the participant selects a whole number (0-10) that best represents the intensity of their pain. The 11-point numerical scale ranges from '0' representing one end of the pain spectrum (e.g. 'no pain') to '10' representing the other end (e.g. 'worst imaginable pain').
Quality of recovery 15 scale | 24 hours after surgery
  Postoperative Quality of Recovery 15 in Turkish scale
Postoperative nausea and vomiting | 24 hours
  Postoperative nausea and vomiting (PONV):
  During follow-up, patients who experience nausea or vomiting will be evaluated using a verbal descriptive PONV scale (0=None, 1=Mild nausea, 2=Moderate nausea, 3=Single episode of vomiting, 4=More than one episode of vomiting).

CONTACTS AND LOCATIONS:
Locations (1):
- Samsun University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.